CLINICAL TRIAL: NCT07313345
Title: Predicting the Pain Outcome of Surgery for Endometriosis
Acronym: PrePOSE
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Endometriosis UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: PrePOSE
Record Dates: First submitted 2025-11-20; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis
Keywords: pelvic pain; fMRI; PROMs
MeSH Terms: conditions — Endometriosis; Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, peritoneal fluid, peritoneum, endometriosis samples (ectopic endometrium and endometrioma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PrePOSE cohort: Women aged 18 - 50 years, with stage III or IV endometriosis, reporting pelvic pain of ≥4/10 and planned for surgical treatment of their endometriosis
  Interventions: Procedure: Surgical treatment of endometriosis

INTERVENTIONS:
Procedure: Surgical treatment of endometriosis — This is an observational study and thus the surgery performed is part of standard clinical care. The procedure will be at the discretion of the operating surgeon/endometriosis multi-disciplinary team and may include bowel resection, stoma formation, ureteric stenting/reimplantation, salpingectomy, oophorectomy or hysterectomy in addition to excision/ablation of endometriosis lesions. Information about the surgical procedure will be collected, but no planned surgical procedure will be an exclusion.

SUMMARY:
This study aims to determine whether the investigators can predict who will get benefit in terms of their pain from surgery for more severe forms of endometriosis. The investigators will use brain imaging to explore this, as it allows meaningful results from a smaller sample of people than if questionnaires alone were relied on.

DETAILED DESCRIPTION:
Endometriosis is a chronic gynaecological condition that affects around 10% of women of reproductive age. This condition can cause debilitating pain, infertility, and poor quality of life. Endometriosis is a condition where tissue resembling the womb lining is present outside of the womb and is associated with an inflammatory pelvic environment. Symptoms of endometriosis can consist of pain during periods, chronic (non-cyclical) pelvic pain, pain during sex, pain when urinating, pain when defecating, and fatigue. Current treatments for endometriosis consist of hormonal, anti-inflammatory and / or analgesic medications and surgery, which is usually laparoscopic ("key-hole"). However, surgery does not always result in a reduction in pain for patients with endometriosis, therefore, it is important to try and understand which patients are most likely to benefit from surgery for their pain management.

Endometriosis is categorized into 4 stages (I - IV), ranging from small areas of tissue that do not extend deeply (stage I) to deep lesions associated with significant scarring of the pelvis and ovarian cysts (endometriomas). Interestingly, symptoms do not correlate with stage of disease. An NIHR funded clinical trial is currently investigating whether surgical treatment of superficial peritoneal endometriosis is of clinical benefit (ESPriT2) and is expected to report early in 2026 (recruitment and baseline data collection are complete). However, women with more severe forms of the disease are excluded from this trial. Surgery is commonly recommended for those with more extensive disease (stages III and IV), however, the risks of surgery are considerably greater for these patients including risk of bladder and bowel damage (sometimes requiring stoma formation) and a negative impact on future fertility. Therefore it is important to better understand who will benefit from this type of surgery. Rather than performing a full clinical trial, the investigators will use a set of experimental tests that allow pain to be understood in more detail meaning less people need to be included in the study and results will be available sooner.

In the present study, patients with pelvic endometriosis at stage III or IV with planned surgical treatment scheduled will be recruited to the project. Participants taking part will provide data at 5 different time points: Time point 1 will consist of several baseline questionnaires, an experimental sensory assessment, and a brain functional magnetic resonance imaging (fMRI) scan. Time point 2 will be the date of their endometriosis surgery, where a questionnaire will be taken, the surgery will be completed, and several biological samples (e.g. blood and small amounts of pelvic fluid and tissue) will be taken. Time points 3 (3 months post-surgery), 4 (6 months post-surgery), and 5 (12 months post-surgery) will consist of completing online questionnaires. All data collected within this project will be used to investigate pain outcome following endometriosis surgery. This research is funded by NIHR BRC.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to give informed consent
* aged between 18 and 50 years of age
* female or born female
* diagnosed with stage III or IV endometriosis by scan (MRI or USS) or previous surgery
* surgical treatment of severe endometriosis planned (surgical procedure at discretion of operating surgeon)
* reports pelvic pain of ≥4/10 (measured using a 0 - 10 numerical rating scale asking about the participant's worst pelvic pain associated with their endometriosis)
* reasonably fluent in English
* in the Investigator's opinion, is able and willing to comply with all study requirements
* willing to allow his or her General Practitioner and consultant to be notified of participation in the study

Exclusion Criteria:

* pregnant, lactating or planning pregnancy during the course of the study
* contraindication to MRI

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients on the waiting list for surgery for severe endometriosis at the Oxford University Hospitals NHS Trust
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Brain response to punctate stimulation of the calf | prior to surgery
  BOLD (Blood oxygen level dependent) response measured with fMRI. Analysis will determine whether BOLD response prior to surgery can predict the pain response (at 12 months post-surgery) to surgical treatment of severe endometriosis.

SECONDARY OUTCOMES:
Brain connectivity at rest | prior to surgery
  Resting state connectivity measured with fMRI
Brain volume | prior to surgery
  Brain volume measured with MRI
Non-cyclical pelvic pain measured on an 11 point numerical rating scale (NRS) | prior to surgery and at 12 months post-surgery
  NRS anchored with 0=no pain, 10=worst pain imaginable
Pain widespreadness | Prior to surgery
  Measured with the Michigan Body Map. The higher the score the more widespread the pain.
Neuropathic-like pain | prior to surgery
  Measured with the painDETECT scale. Scores range from -1 to 38. Higher scores represent more likely to have a neuropathic component to pain.
Pain catastrophising | Prior to surgery
  Measured with the pain catastrophising scale (Sullivan). Scores range from 0 - 52 with high scores representing higher levels of pain catastrophising. Although three sub scales exist they will not be assessed for the purposes of these main analyses.
Pain self-efficacy | Prior to surgery
  Measured with the pain self-efficacy scale. Scores range from 0 to 60, with higher scores indicating greater confidence in managing pain.
Expectation of surgical efficacy | Prior to surgery
  Measured on an 8 point verbal rating scale anchored with 0=I do not suffer from this and do not expect that will change, 1=very marked improvement, 2=marked improvement, 3=minimal improvement, 4=no change, 5=minimal worsening, 6=marked worsening, 7=very marked worsening

OTHER OUTCOMES:
Quantitative Sensory Testing (QST) of the lower abdomen and left hand according to the German Neuropathic Pain Network Protocol | Prior to surgery
  Individual measures and the overall sensory profile cluster (derived according to Vollert)

CONTACTS AND LOCATIONS:
Overall Officials: Katy Vincent, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospitals Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Once data analysis is complete all data will be deposited in appropriate publicly accessible repositories as required by the funders. No personal data will be included in these datasets.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of all manuscripts from the study
Access Criteria: Data will be publicly accessible